CLINICAL TRIAL: NCT04129983
Title: Prospective Study of Sudden Deafness
Brief Title: Treatment of Sudden Deafness With Prednisone+Hyperbaric Oxygen and Prednisone+Somatosensory Stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dan Su (Other)
Responsible Party: Sponsor-Investigator, Dan Su, principal investigator, The First Affiliated Hospital of Anhui Medical University
Organization: The First Affiliated Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pssd
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hearing Loss, Sudden; Prednisone Acetate; Hyperbaric Oxygen; Somatic Stimulus
Keywords: Hearing Loss, Sudden; Prednisone acetate; Hyperbaric oxygen; Somatic stimulus
MeSH Terms: conditions — Hearing Loss, Sudden | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisone acetate + somatosensory stimulation (Experimental): Prednisone acetate 1 mg/kg body weight * 7 days and somatosensory stimulation 30 days were given to sudden deafness patients.
  Interventions: Combination Product: Drugs and Stimulation
- Prednisone acetate + hyperbaric oxygen (Experimental): Prednisone acetate 1mg / kg body weight * 7 days and hyperbaric oxygen 15 days were given to sudden deafness patients.
  Interventions: Combination Product: Drugs and Stimulation

INTERVENTIONS:
Combination Product: Drugs and Stimulation — 60 cases of sudden deafness were inquired about their medical history and examined by hearing and cranial magnetic resonance. They were randomly divided into two groups and given different treatments. The hearing test was repeated every 7 days. One month and three months after the treatment, the hearing examination was reexamined.

SUMMARY:
To study the effective treatment of sudden deafness by giving prednisone, hyperbaric oxygen and somatosensory stimulation to sudden deafness patients.

DETAILED DESCRIPTION:
60 cases of sudden deafness within 2 months of 14-80 years old were randomly divided into two groups. They underwent hearing tests, magnetic resonance imaging of the head, and routine hospital admissions. One group was given prednisone for 1 mg / kg body weight × 7 days + somatosensory stimulation × 30 days, the other group was given prednisone for 1 mg / kg body weight × 7 days + hyperbaric oxygen × 15 days, and repeated electrical audiometry every week. One month and three months after the experiment, repeated audiometry.

ELIGIBILITY:
Inclusion Criteria:

* Sudden deafness
* History within 2 months
* Age 14-80

Exclusion Criteria:

* Neurological diseases (such as brain tumors)
* Patients with mental / mental illness undergoing treatment
* Pregnant women and patients with other untreatable diseases
* Finding the cause of sensorineural deafness
* Patients Not Suitable for Hyperbaric Oxygen
* A patient with dermatosis

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Audiometry | Three months from the patient's selection to the end of treatment
  Evaluate the patient's hearing to determine whether it has improved.
Cranial magnetic resonance imaging | When patients are enrolled
  Judging whether the patient's inner ear has pathological changes or not

CONTACTS AND LOCATIONS:
Overall Officials: Busheng Tong, doctor, Study Director — E.N.T. department of the First Affiliated hospital of Anhui Medical University
Locations (1):
- E.N.T. department of the First Affiliated hospital of Anhui Medical University, Hefei, Anhui, China